CLINICAL TRIAL: NCT01072331
Title: Pharmacokinetic/Pharmacodynamic Study of MP-513 in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: Pharmacokinetic/Pharmacodynamic Study of MP-513 With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3000-A12
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MP-513 10 mg, once a day, for 4 weeks (Experimental)
  Interventions: Drug: MP-513
- MP-513 20 mg, once a day, for 4 weeks (Experimental)
  Interventions: Drug: MP-513
- Placebo of MP-513 (Placebo Comparator)
  Interventions: Drug: Placebo of MP-513

INTERVENTIONS:
Drug: MP-513 — MP-513 10 mg, once a day, for 4 weeks
  Arms: MP-513 10 mg, once a day, for 4 weeks
Drug: MP-513 — MP-513 20 mg, once a day, for 4 weeks
  Arms: MP-513 20 mg, once a day, for 4 weeks
Drug: Placebo of MP-513 — MP-513 placebo, once a day, for 4 weeks
  Arms: Placebo of MP-513

SUMMARY:
The purpose of this study is to evaluate the effect of MP-513 on 24-h glycemic control in patients with type 2 Diabetes for 4 weeks administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 20 - 75 years old
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 8 weeks before administration of investigational drug
* Patients whose HbA1c is ≥6.5% and <10.0%
* Patients who were not administered diabetes therapeutic drugs prohibited for concomitant use within 8 weeks before administration of investigational drug.

Exclusion Criteria:

* Patients with type 1 diabetes, diabetes mellitus caused by pancreas impairment, or secondary diabetes (Cushing disease, acromegaly, etc)
* Patients who are accepting treatments of arrhythmias
* Patients with serious diabetic complications
* Patients who are the excessive alcohol addicts
* Patients with severe hepatic disorder or severe renal disorder.
* Patients who are pregnant, lactating, and probably pregnant patients, and patients who can not agree to contraception

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation; Tadashi Yoshida, MD, Study Director — Tanabe Pharma Corporation
Locations (1):
- Suita, Osaka, Japan

REFERENCES:
- [Result] Eto T, Inoue S, Kadowaki T. Effects of once-daily teneligliptin on 24-h blood glucose control and safety in Japanese patients with type 2 diabetes mellitus: a 4-week, randomized, double-blind, placebo-controlled trial. Diabetes Obes Metab. 2012 Nov;14(11):1040-6. doi: 10.1111/j.1463-1326.2012.01662.x. Epub 2012 Jul 29. PMID 22776014

RESULTS

PARTICIPANT FLOW:
Groups:
- MP-513 10 mg: MP-513 10 mg once a day for 4 weeks
- MP-513 20 mg: MP-513 20 mg once a day for 4 weeks
- Placebo of MP-513: Placebo of MP-513 a day for 4 weeks
Period: Overall Study
Arm/Group | MP-513 10 mg | MP-513 20 mg | Placebo of MP-513
Started | 34 | 33 | 32
Completed | 34 | 33 | 32
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP-513 10 mg | MP-513 20 mg | Placebo of MP-513 | Total
Number analyzed (Participants) | 34 | 33 | 32 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (11.5) | 57.1 (8.7) | 58.6 (8.9) | 57.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 6 | 15
  Male | 29 | 29 | 26 | 84

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 2-h Postprandial Glucose (Breakfast, Lunch and Dinner)
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Arm/Group | MP-513 10 mg | MP-513 20 mg | Placebo of MP-513
Number analyzed (Participants) | 34 | 33 | 32
mg / dL
  2-h Postprandial Glucose (breakfast) | -56.2 (5.5) | -43.7 (5.8) | -5.5 (6.0)
  2-h Postprandial Glucose (lunch) | -43.1 (6.5) | -36.9 (7.0) | -8.3 (7.0)
  2-h Postprandial Glucose (dinner) | -41.8 (5.4) | -40.5 (5.7) | -4.3 (5.8)

2. Secondary Outcome: Change From Baseline in 24-h Mean Glucose
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Arm/Group | MP-513 10 mg | MP-513 20 mg | Placebo of MP-513
Number analyzed (Participants) | 34 | 33 | 32
mg / dL | -34.722 (3.885) | -30.921 (4.005) | -5.402 (4.037)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Arm/Group | MP-513 10 mg | MP-513 20 mg | Placebo of MP-513
Number analyzed (Participants) | 34 | 33 | 32
mg / dL | -20.7 (2.7) | -20.5 (2.8) | -6.9 (2.8)

4. Primary Outcome: Change From Baseline in Plasma Glucose Area Under the Curve (AUC) 0 to 2h (Breakfast, Lunch and Dinner)
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: mg・h / dL
Arm/Group | MP-513 10 mg | MP-513 20 mg | Placebo of MP-513
Number analyzed (Participants) | 34 | 33 | 32
mg・h / dL
  Plasma Glucose AUC (breakfast) | -82.114 (8.028) | -75.437 (8.321) | -8.950 (8.294)
  Plasma Glucose AUC (lunch) | -92.947 (10.592) | -86.843 (11.328) | -6.884 (11.184)
  Plasma Glucose AUC (dinner) | -75.204 (9.660) | -85.192 (10.158) | -11.271 (10.218)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | MP-513 10 mg | MP-513 20 mg | Placebo of MP-513
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 8/34 | 6/33 | 9/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP-513 10 mg (N=34) | MP-513 20 mg (N=33) | Placebo of MP-513 (N=32)
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 1
Glucose urine present (Investigations) | 1 | 0 | 3
Blood urine present (Investigations) | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other